CLINICAL TRIAL: NCT02550925
Title: A Novel Acceptance-Based Intervention for Anxious Cancer Survivors
Brief Title: Acceptance and Commitment Therapy (ACT) for Anxious Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: American Cancer Society, Inc. (Other); Rocky Mountain Cancer Centers (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Joanna Arch, Associate Professor, Department of Psychology and Neuroscience, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RSG-15-020-01
Record Dates: First submitted 2015-07-30; First posted 2015-09-16 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: Cancer survivors
MeSH Terms: conditions — Neoplasms | interventions — Population Groups

STUDY DESIGN:
Masking Description: Note: 139 individuals enrolled. 4 dropped out after consent, before baseline data collection, leaving 135 individuals with data.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment Therapy Group (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) Group
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) Group — A 7-session Acceptance and Commitment Therapy (ACT) group intervention
  Arms: Acceptance and Commitment Therapy Group
Behavioral: Usual Care — Check in with clinical social worker at oncology care site and obtain list of supportive resources
  Arms: Usual Care

SUMMARY:
This randomized clinical trial compares group acceptance and commitment therapy (ACT) to usual care for cancer survivors experiencing anxiety following the end of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults in the Greater Boulder/ Denver, Colorado area who had cancer and completed primary cancer treatment (surgery, chemotherapy, and/or radiation) within the previous 18 months
2. For solid tumor cancers: Show no current evidence of disease for solid-tumor cancers (of any cancer type or initial stage). For lymphoproliferative disorders such as chronic lymphocytic leukemia and indolent non-Hodgkin's lymphoma: In remission or asymptomatic after initial treatment and are followed with active surveillance.
3. Screen positive for anxiety symptoms on the study screener
4. Able to speak, read, and write English fluently
5. Willing and able to participate in an ACT group once a week for 7 weeks
6. Willing and able to complete online questionnaires and phone interviews at designated assessment points

Exclusion Criteria:

1. Current moderate to high suicide risk
2. History of chronic untreated trauma (unrelated to their cancer)
3. Psychiatric hospitalization or suicide attempt in the past 5 years

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms | Baseline to Post and (3- and 6-month) Follow Up
  Method of assessment: questionnaire

SECONDARY OUTCOMES:
Depressive symptoms | Baseline to Post and (3- and 6-month) Follow Up
  Method of assessment: questionnaire
Medical resource use | Baseline to Post and (3- and 6-month) Follow Up
  Method of assessment: survey of medical care use
Fear of cancer recurrence | Baseline to Post and (3- and 6-month) Follow Up
  Method of assessment: questionnaire
Sense of life meaning | Baseline to Post and (3- and 6-month) Follow Up
  Method of assessment: questionnaire
Fatigue / Vitality | Baseline to Post and (3- and 6-month) Follow Up
  Method of assessment: questionnaire
Anxiety disorder severity | Baseline to Post and 6-month Follow Up
  Method of assessment: diagnostic interview

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

REFERENCES:
- [Background] Arch JJ, Mitchell JL. An Acceptance and Commitment Therapy (ACT) group intervention for cancer survivors experiencing anxiety at re-entry. Psychooncology. 2016 May;25(5):610-5. doi: 10.1002/pon.3890. Epub 2015 Jun 29. No abstract available. PMID 26130586
- [Derived] Arch JJ, Mitchell JL, Genung SR, Judd CM, Andorsky DJ, Bricker JB, Stanton AL. Randomized trial of acceptance and commitment therapy for anxious cancer survivors in community clinics: Outcomes and moderators. J Consult Clin Psychol. 2021 Apr;89(4):327-340. doi: 10.1037/ccp0000630. PMID 34014694
- [Derived] Arch JJ, Mitchell JL, Genung SR, Fisher R, Andorsky DJ, Stanton AL. A randomized controlled trial of a group acceptance-based intervention for cancer survivors experiencing anxiety at re-entry ('Valued Living'): study protocol. BMC Cancer. 2019 Jan 18;19(1):89. doi: 10.1186/s12885-019-5289-x. PMID 30658621